CLINICAL TRIAL: NCT03389568
Title: The Effects of Singing-based Music Therapy Program on the Level of Psychoemotional Benefits in Caregivers of ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0963
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Primary Family Caregivers of ICU Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention for caregivers of ICU patients (Experimental)
  Interventions: Behavioral: singing-based music therapy program

INTERVENTIONS:
Behavioral: singing-based music therapy program — A single 1-hour singing-based intervention is conducted with each primary caregiver of an ICU patient. The intervention is composed of three steps: 1) listening to a participant's preferred music and identifying his and her emotional states (15 minutes), (2) singing for emotional changes (30 minutes), and (3) discussing what he or she experiences during singing and identifying how they apply such experience to their personal use of music for emotional changes in his or her everyday life (15 minutes).

SUMMARY:
This study applies an one-group pre-posttest design. Primary family caregivers of ICU patients are recruited. After obtaining an informed consent form from each participant, he or she participates in an individual 1-hour singing-based music therapy intervention. At pre- and posttest, the changes in the level of depression, anxiety, and emotional states are measured.

DETAILED DESCRIPTION:
* Background: Family caregivers of ICU patients experience high level of distress due to the severity of illness that their family members demonstrate and the perceived limitation in control during their caregiving. This psychological issue in family caregivers have been documented to affect not only the caregivers' psychosocial health but also the quality of care for patients, which would also be influencing factors for treatment outcomes of patients. As such, family-centered care has been emphasized in related professions. Intervention efforts for family caregivers are also of interest. Given that music has been evidenced to effectively alleviate emotional stress of caregivers and that musical activities can be used in an individualized way at different levels, the use of music for addressing psychosocial needs of this population is potential. Among musical activities, singing is one of the most common activities and also available in everyday life regardless of the level of musical background in the past, which increases the possibility to utilize it as a personal strategy for individuals with a broad range of musical experiences and music use.
* Purpose: This study aimed to examine the changes in the level of depression, anxiety, and emotional states of family caregivers of ICU patients after participation in singing-based music therapy intervention.
* Intervention: Singing-based music therapy program consists of the sequences of the following: (1) listening to a participant's preferred music and identifying his and her emotional states, (2) singing for emotional changes, and (3) discussing what he or she experiences during singing and identifying how they apply such experience to their personal use of music for emotional changes in his or her everyday life.
* Measures: In order to examine the changes in the perceived psychological health after participation in singing-based intervention, Center for Epidemiologic Studies Depression Scale (CES-D), State Anxiety Inventory (STAI), and a 100mm visual analog scale for ratings on emotional state are administered. Also, in order to identify and control the effect of level of caregiving burden on current emotional states, Subjective Caregiving Burden Scale is administered.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and over
* Family members (spouse, parents, or children) of patients who stay in the ICU for more than 3 days
* Provision of the majority of unpaid physical, emotional, and/or instrumental care to the patients
* Voluntarily agreement with participation in the study

Exclusion Criteria:

* A history of cognitive impairment (e.g., dementia), psychiatric disorders or neurological disorders
* Indication of discernible hearing deficits
* Difficulties in verbal communication
* If the caregiver's relationship to a patient is close friend or relatives (not immediate family of patients)
* Refusal to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | 5 minutes before the intervention
  This study aimed to examine the changes in the measured CES-D in caregivers of ICU patients after participation in music therapy intervention. CES-D is the self-administered scale and consists of Likert-type 20 items on depressed affect, positive affect, somatic activity, and interpersonal relationship. The value measured from this scale indicates a level of depressive symptoms.
Center for Epidemiologic Studies Depression Scale (CES-D) | 5 minutes after the intervention
  This study aimed to examine the changes in the measured CES-D in caregivers of ICU patients after participation in music therapy intervention. CES-D is the self-administered scale and consists of Likert-type 20 items on depressed affect, positive affect, somatic activity, and interpersonal relationship. The value measured from this scale indicates a level of depressive symptoms.

SECONDARY OUTCOMES:
State Anxiety Inventory (STAI) for anxiety | 5 minutes before the intervention
  As the secondary outcomes of intervention, changes in the level of anxiety are measured. The level of anxiety is measured by scores on State Anxiety Inventory (STAI). STAI is the self-administered scale and consists of 4-Likert type of 20 items on the perceived emotions in terms of anxiety.
State Anxiety Inventory (STAI) for anxiety | 5 minutes after the intervention
  As the secondary outcomes of intervention, changes in the level of anxiety are measured. The level of anxiety is measured by scores on State Anxiety Inventory (STAI). STAI is the self-administered scale and consists of 4-Likert type of 20 items on the perceived emotions in terms of anxiety.
VAS(Visual Analog Scale) for emotional state | 5 minutes before the intervention
  As the secondary outcomes of intervention, changes in the level of emotional states are measured. For emotional states, a 100mm visual analog scale (VAS) is used for participants to rate how they feel happiness, sadness, anger, fear, and comfort.
VAS(Visual Analog Scale) for emotional state | 5 minutes after the intervention
  As the secondary outcomes of intervention, changes in the level of emotional states are measured. For emotional states, a 100mm visual analog scale (VAS) is used for participants to rate how they feel happiness, sadness, anger, fear, and comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McAdam JL, Dracup KA, White DB, Fontaine DK, Puntillo KA. Symptom experiences of family members of intensive care unit patients at high risk for dying. Crit Care Med. 2010 Apr;38(4):1078-85. doi: 10.1097/CCM.0b013e3181cf6d94. PMID 20124890
- [Result] Melnyk BM, Alpert-Gillis L, Feinstein NF, Crean HF, Johnson J, Fairbanks E, Small L, Rubenstein J, Slota M, Corbo-Richert B. Creating opportunities for parent empowerment: program effects on the mental health/coping outcomes of critically ill young children and their mothers. Pediatrics. 2004 Jun;113(6):e597-607. doi: 10.1542/peds.113.6.e597. PMID 15173543
- [Result] O'Kelly J. Saying it in song: music therapy as a carer support intervention. Int J Palliat Nurs. 2008 Jun;14(6):281-6. doi: 10.12968/ijpn.2008.14.6.30023. PMID 18928132